CLINICAL TRIAL: NCT00743912
Title: A Phase 1, Single Arm, Open-Label Study to Evaluate the Effect of Rifaximin 550 MG Tablets TID on the Pharmacokinetics of Orally Administered Midazolam in Healthy Male and Female Volunteers
Brief Title: Open-Label Study to Evaluate the Effect of Rifaximin on Midazolam in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RFDI1008
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Pharmacokinetic
Keywords: rifaximin; midazolam; pharmacokinetics
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): open-label rifaximin 550 mg TID
  Interventions: Drug: rifaximin

INTERVENTIONS:
Drug: rifaximin — 550 mg TID

SUMMARY:
The primary objective of this study is to determine if rifaximin, administered daily has an effect on the cytochrome P450 (CYP) isoenzyme 3A4, by examining any changes in the pharmacokinetics of midazolam (a CYP3A4 substrate), when co-administered.

DETAILED DESCRIPTION:
This is a single-site, single-arm, open-label, drug-interaction study that examines the effect of rifaximin (RFX), 550 mg 3 times daily (TID; 1650 mg/day), on orally administered (PO) midazolam (MDZ) 2 mg (administered as a 2 mg dose in 1 mL of midazolam HCL Syrup; 2 mg/mL) when dosed for 7 and 14 consecutive days, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patient is medically normal
* Patient has normal laboratory values
* Patient has the ability to understand the requirements of the study

Exclusion Criteria:

* HIV
* Hepatitis B
* Hepatitis C
* History of renal, hepatic, endocrine, oncological, gastrointestinal or cardiovascular disease.
* History of epilepsy, asthma, diabetes, psychosis, glaucoma or severe head injury.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Individual midazolam and rifaximin plasma concentrations and pharmacokinetic parameters will be summarized. | 21 to 38 days (including a 21 day screening period)

SECONDARY OUTCOMES:
Overall safety assessments will include the incidence, intensity, and type of adverse events, and clinically significant changes in the patient's physical examination, vital signs and laboratory results. | 21 tyo 38 days

CONTACTS AND LOCATIONS:
Overall Officials: William Lewis, MD, Principal Investigator — Covance CRU, Inc